CLINICAL TRIAL: NCT05052827
Title: Anabolic Potential of Dairy and Dairy Proteins for Active Children and Adolescents
Brief Title: Determining the Effect of Protein Quality on Post-exercise Anabolism in Active Youth
Acronym: PQS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 36378
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Dietary Proteins
Keywords: protein quality; growth; indicator amino acid oxidation; children; adolescent
MeSH Terms: interventions — Soybean Proteins

STUDY DESIGN:
Intervention Model Description: Using a single-blind randomized counterbalanced crossover design, participants will complete three metabolic trials providing 0.35 g/kg FFM of either milk protein concentrate (MPC), rice protein isolate (RPI), or soy protein isolate (SPI) following a bout of variable intensity exercise.
Who Masked: Participant
Masking Description: As the study was a single-blind crossover design, the randomization of the protein type will be blinded to the participants only. The allocation concealment in relation to the liquid meal will be done by providing the same relative protein content (0.35 g/kg FFM) within the same volume of fluid, (8 ml/kg) to match the exercise-induced fluid loses, in opaque bottles. Additional carbohydrate (0.4g/kg) and artificial sweetener will be added to improve the organoleptic properties of the beverages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Children (Active Comparator): Participants underwent 3 metabolic trials in a randomized crossover fashion, where they were provided with an isonitrogenous quantities of either milk protein concentrate, soy protein isolate, and rice protein isolate following a standardized bout of variable intensity exercise.
  Interventions: Dietary Supplement: Milk Protein Concentrate; Dietary Supplement: Rice Protein Isolate; Dietary Supplement: Soy Protein Isolate
- Adolescent Females (Active Comparator): Participants underwent 3 metabolic trials in a randomized crossover fashion, where they were provided with an isonitrogenous quantities of either milk protein concentrate, soy protein isolate, and rice protein isolate following a standardized bout of variable intensity exercise.
  Interventions: Dietary Supplement: Milk Protein Concentrate; Dietary Supplement: Rice Protein Isolate; Dietary Supplement: Soy Protein Isolate
- Adolescent Males (Active Comparator): Participants underwent 3 metabolic trials in a randomized crossover fashion, where they were provided with an isonitrogenous quantities of either milk protein concentrate, soy protein isolate, and rice protein isolate following a standardized bout of variable intensity exercise.
  Interventions: Dietary Supplement: Milk Protein Concentrate; Dietary Supplement: Rice Protein Isolate; Dietary Supplement: Soy Protein Isolate

INTERVENTIONS:
Dietary Supplement: Milk Protein Concentrate — Protein provided at 0.35 g/kg fat free-mass. Macronutrient and Amino Acid Content provided below.
  Per 100 g protein powder:
  Calories (Cal): 363 Carbs (g): 5.60 Protein (g): 82.60 Fat (g): 1.12 Total BCAA (g): 15.67 Total EAA (g): 34.66 Total AA (g): 83.27
  Other Names: MPC, Idaho Milk Products (Grade A)
Dietary Supplement: Rice Protein Isolate — Protein provided at 0.35 g/kg fat free-mass. Macronutrient and Amino Acid Content provided below.
  Per 100 g protein powder:
  Calories (Cal): 394 Carbs (g): 6.50 Protein (g): 86.70 Fat (g): 2.39 Total BCAA (g): 14.98 Total EAA (g): 30.62 Total AA (g): 86.11
  Other Names: RPI, Axiom Foods - Organic Oryzatein Silk 90
Dietary Supplement: Soy Protein Isolate — Protein provided at 0.35 g/kg fat free-mass. Macronutrient and Amino Acid Content provided below.
  Per 100 g protein powder:
  Calories (Cal): 377 Carbs (g): 2.12 Protein (g): 88.8 Fat (g): 0.60 Total BCAA (g): 13.88 Total EAA (g): 31.74 Total AA (g): 89.39
  Other Names: MyProtein - Soy Protein Isolate

SUMMARY:
Leucine-enriched proteins (e.g., dairy) are more effective than plant-based sources for supporting post-exercise rates of muscle protein synthesis in adults. However, the impact of protein quality on protein synthesis and acute markers of growth in active children are unknown. Using a randomized crossover design, the investigators will compare the effects of ingesting 0.35g/kg fat free mass (FFM) of either milk protein concentrate (MPC), rice protein isolate (RPI), or soy protein isolate (SPI) following a bout of variable intensity exercise with whole-body protein kinetics (i.e., oxidation, synthesis, breakdown, and net balance) determined by oral [13C]phenylalanine tracer methodology.

DETAILED DESCRIPTION:
In adults, dairy protein is more effective than non-dairy sources at supporting recovery from exercise; however, it is not well understood if protein quality impacts short-term markers of growth in the same manner in active youth. Therefore, it is essential to understand whether different anabolic responses to varying protein quality persist in children, in order to maximize lean tissue accretion specifically during these periods of exponential growth. Thus, assessing the impact of protein quality on post-exercise protein synthesis and whole-body protein balance in active children would help provide valuable maturation-specific nutritional information. Moreover, these studies investigating the effects of protein quality in adults required the use of invasive techniques (i.e., muscle biopsies and indwelling catheters for blood draws) and are not suitable for vulnerable populations like children. As a result, the study of protein quality in children requires non-invasive alternative approaches and novel methods to advance our understanding of the nutritional best practices for active youth.

The overall objective of this investigation is to examine the impact of protein quality on post-exercise protein synthesis and acute markers of "growth" (i.e., net protein balance) in active youth (children and adolescents). Using the minimally invasive indicator amino acid oxidation (IAAO) methodology, we will determine the ability of milk, rice, and soy proteins to support whole-body protein synthesis and net-protein balance during recovery from an acute bout of sport specific moderate-to-vigorous physical activity.

The primary aim of the present study is to compare the ability of dairy and non-dairy alternatives (i.e., plant-based protein sources) to support post-exercise protein synthesis and net-protein balance in active, growing youth. The investigators hypothesize that the ingestion of milk protein concentrate (MPC) will result in a lower indicator amino acid oxidation (i.e., greatest protein synthesis) and higher net protein balance after exercise in both children and adolescents, compared to an isonitrogenous (i.e., equal protein amount) quantity of soy (SPI) and rice (RPI) protein isolate. This is predicated on the relative deficiency of branched-chain amino acids (BCAA) and other essential amino acids (EAA), specifically lysine and methionine, in RPI and SPI respectively, compared to MPC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy will be defined as screened by the PAR-Q+ (The Physical Activity Readiness Questionnaire for everyone)
* Regularly active, as defined by being in the top 20% of age specific scores on the iPAQ (the International Physical Activity Questionnaire)
* Between the ages of 8 to 16 years
* An age and sex-specific minimum of 75th percentile Beep Test level

Exclusion Criteria:

* Inability to meet health and physical activity guidelines according to the PAR-Q+ and iPAQ
* Inability to adhere to any of the protocol guidelines
* Biological age outside of -0.5 to +1.5 years from PHV for adolescents, and > -1 years from PHV for children

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
F13CO2 | The rate of 13CO2 excretion based upon baseline (t=30 minutes) and isotopic steady state (t=360-420 minutes) 13CO2 enrichments in the breath and resting VCO2
  Rate of 13CO2 excretion

SECONDARY OUTCOMES:
Whole-Body Phenylalanine Kinetics | Whole-Body Net Protein Balance will be calculated based upon baseline (t=30 minutes) and isotopic steady state (t=360-420 minutes) 13CO2 enrichments in the breath and 1-[13C]phenylalanine enrichments in the urine
  Whole-Body Net Protein Balance

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, PhD, Principal Investigator — University of Toronto; Hugo JW Fung, MSc, Study Director — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No